CLINICAL TRIAL: NCT05678244
Title: Intravenous Acetaminophen For Postoperative Pain in the Neonatal Intensive Care Unit: A Feasibility Randomized Controlled Trial
Brief Title: Intravenous Acetaminophen For Postoperative Pain in the Neonatal Intensive Care Unit
Acronym: IVA POP NICU
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: McMaster Children's Hospital (Other)
Responsible Party: Principal Investigator, Victoria Archer, Resident Principal Investigator, McMaster Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14887-GRA
Record Dates: First submitted 2022-12-06; First posted 2023-01-10 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Pain, Postoperative; Pain
Keywords: acetaminophen; pain; neonate; infant; tylenol; paracetamol; postoperative; surgery
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Acetaminophen

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to the control or comparator group. There will be 60 patients enrolled, with 30 patients per arm.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: IV acetaminophen and saline appear identical in solution. They will be administered at identical rates. Care providers, participants' parents, investigators, outcomes assessors, and statisticians will remain blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Comparator (Active Comparator): Standard of care + IV acetaminophen:
  Baseline fentanyl infusion, with dosage escalations, deescalations, and additional boluses and analgesics (excluding oral or rectal acetaminophen) determined by the patient's physician (this represents standard of care at this institution) with the addition of IV acetaminophen every 4 or 6 hours at weight-appropriate doses based on the patient's gestational age.
  Interventions: Drug: Acetaminophen
- Placebo (Placebo Comparator): Standard of care + placebo:
  Baseline fentanyl infusion, with dosage escalations, deescalations, and additional boluses and analgesics (excluding oral or rectal acetaminophen) determined by the patient's physician (this represents standard of care at this institution) with the addition of an IV saline placebo every 4 or 6 hours at a rate which would mimic their dose of acetaminophen.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acetaminophen — IV acetaminophen will be added to standard of care opioid based pain regimes.
  Arms: Comparator
Drug: Placebo — In control group placebo will be added to standard of care opioid based pain regimes.
  Arms: Placebo

SUMMARY:
The goal of this pilot randomized clinical trial is to determine the effect of the addition of IV acetaminophen to opioid-based pain regimes for infants admitted to the neonatal intensive care unit (NICU) after surgery.

This is a pilot trial; the main goals are to make sure our study methods work before performing a larger study.

The main clinical aims are:

1. Determine if adding IV acetaminophen reduces pain
2. Determine if adding IV acetaminophen reduces opioid use
3. Determine if adding IV acetaminophen reduces complications

Participants will be randomized to two groups:

Comparator: Fentanyl and IV acetaminophen Control: Fentanyl and placebo

Patients will receive either IV acetaminophen or placebo at regular intervals for seven days after surgery. Patients will be followed daily during that period. Charts will be reviewed at 90-days for final outcomes.

DETAILED DESCRIPTION:
Purpose: Opioid use in neonates is associated with short and long-term adverse events. Multi-modal pain control offers the ability to control pain while reducing opioid exposure. This topic has been relatively unexamined in preterm and term neonates. Specifically, this trial aims to evaluate the effect of adding IV acetaminophen to standard opioid-based pain regimes in neonates in the neonatal intensive care unit (NICU) undergoing major abdominal and thoracic surgery.

Objectives: The primary aim of the proposed study is to determine the feasibility and cost of conducting a multicenter, randomized control trial to compare the efficacy of IV acetaminophen and fentanyl, to fentanyl and saline placebo, in terms of reduction of postoperative pain, opioid use, adverse events. The primary outcome is feasibility; secondarily, efficacy and safety will be assessed.

Design: This single-center, parallel-arm, placebo-controlled, fully blinded, randomized controlled external feasibility trial will enroll patients admitted in the neonatal intensive care unit (NICU) who have undergone major, thoracic, or abdominal surgery. Patients will be randomized 1:1, with parallel allocation to receive acetaminophen and fentanyl or fentanyl and saline placebo. All study staff, clinical staff and guardians will be blinded. As this is a pilot study, no sample size will be calculated, however; we aim to enroll 60 patients. A sample size calculation will be completed for the full RCT if it is deemed feasible from the results of this study. Patients will be followed for the day of surgery and the following 7 postoperative days (192 hours) and have their charts reviewed at 90 days.

Impact: The results of this study will be used to determine the feasibility of conducting a multi-center RCT to assess the effect of IV acetaminophen on fentanyl infusions in postoperative neonatal patients. The effect of IV acetaminophen for postoperative pain in preterm neonates has yet to be studied, this trial would generate novel insights into its efficacy. The prolonged follow-up period would also provide novel insights into recovery throughout the entire perioperative period.

ELIGIBILITY:
Inclusion Criteria:

1. Neonates, admitted to McMaster Children's Hospital NICU
2. Has had major open, thoracic or abdominal surgery (see appendix 1, table 6).
3. Informed consent obtained from guardian(s)

Exclusion Criteria:

1. Hepatic dysfunction

   * AST, ALT or Bilirubin > 3x upper limit of normal
   * INR ≥ 3.0 or PT greater than 20s regardless of vitamin K administration
2. Renal dysfunction

   * Increase in serum creatinine ≥ 2x baseline (baseline: lowest value in first 5 days of hospitalization)
   * Urine output < 0.5 mL/kg/h for ≥ 12h
3. Allergy or intolerance to acetaminophen or fentanyl
4. Acetaminophen administration within 24 hours of the end of surgery
5. Nerve blocks or epidurals
6. Refusal or withdrawal of consent
7. Enrolment in another competing trial
8. No later than 12 hours after the end of surgery
9. 12 months post gestational age or greater in age
10. Birthweight greater or equal to 2,500g.
11. Discharged from the McMaster NICU

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2023-04-17 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | through study completion, an average of 1.5 years
  Mean number of patients randomized per month
Follow up rate | 90 days
  Number of patients followed in completion from postoperative day 0 to 7
Medication compliance | 7 days
  Number of patients who received at least 80% of doses of study drugs at the correct dose and interval
Blinding index | 7 days
  Responses of nurse's physician's, and research staff's guess of group assignment (control vs treatment) compared to actual group assignment

SECONDARY OUTCOMES:
Postoperative Pain | every 6 hours for entire study period (7 days after surgery)
  Measured by the N-PASS Pain Scale as units on the scale (scale ranges from 0-10)
Daily fentanyl consumption | daily for 7 days
  Fentanyl consumption will be recorded for each patient for each 24-hour period in the study period. Will be recorded in mcg/kg.
Total fentanyl consumption | 7 days
  Daily fentanyl consumption will be added together for the entire study period to determine the total amount of fentanyl consumed in mcg/kg.
Daily Consumption of other analgesics | daily for 7 days
  Consumption of other analgesics will be recorded for each patient for each 24-hour period in the study period. Will be recorded in mg or mcg /kg.
Total consumption of other analgesics | 7 days
  Daily consumption of other analgesics will be added together for the entire study period to determine the total amount of fentanyl consumed in mg or mcg/kg.
Invasive ventilation | 90 days
  Length of time requiring intubation
Non-invasive ventilation | 90 days
  Length of time requiring CPAP, BiPAP, or supplemental oxygen
Enteral feeds | 90 days
  Time to first enteral feeds and time to full enteral feeds (using NICU's calculated goal feed)
Bowel movement | 90 days
  Time to first bowel movement
Glycerin suppository use | 90 days
  Number of patients requiring one or more glycerin suppositories
Length of stay | 90 days
  with discharge destination

OTHER OUTCOMES:
Vomiting | 7 days
  Number of patients with ≥ 1 episode of vomiting documented
NG/Vygone | 90 days
  Number of patients, mean duration
Reintubation | 90 days
  Number of patients
Apnea | 7 days
  Number of patients with oxygen saturation less than 94% or RR less than 20 breaths/min for more than 30 seconds
Naloxone administration | 7 days
  Number of patients
Bradycardia | 7 days
  Number of patients with HR less than 100 for more than 30 seconds
Hypotension | 7 days
  Number of patients with SBP less than 60, or requiring vasoactive medication
Foley catheterization | 7 days
  Number of patients, mean duration
Feeding intolerance | 7 days
  Number of patients: feeds stopped or decreased due to vomit/increased gastric output, or if diagnosed by the treating team
Hepatic injury | 90 days
  Number of patients with hepatic injury as defined in the protocol
Mortality | 90 days
  all cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: Mark Walton, MD, Principal Investigator — McMaster University
Locations (1):
- McMaster Children's Hospital, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Archer VA, Samiee-Zafarghandy S, Farrokyhar F, Briatico D, Braga LH, Walton JM. Intravenous acetaminophen for postoperative pain in the neonatal intensive care unit: A protocol for a pilot randomized controlled trial (IVA POP). PLoS One. 2023 Nov 20;18(11):e0294519. doi: 10.1371/journal.pone.0294519. eCollection 2023. PMID 37983228